CLINICAL TRIAL: NCT01426867
Title: A Descriptive Comfort Study of Brinzolamide 1% / Brimonidine Tartrate 0.2% Fixed Combination Ophthalmic Suspension, Brinzolamide 1% Ophthalmic Suspension and Brimonidine Tartrate 0.2% Ophthalmic Solution in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: A Comfort Study of Brinzolamide 1% / Brimonidine 0.2% Fixed Combination, Brinzolamide 1% and Brimonidine 0.2%
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-11-002
Record Dates: First submitted 2011-08-24; First posted 2011-09-01 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension; Intraocular Pressure; Brinzolamide; Brimonidine
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brinz/Brim (Experimental): Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension, 1 drop instilled in each affected eye 3 times a day for 7 days
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
- Brinzolamide (Active Comparator): Brinzolamide ophthalmic suspension, 1%, 1 drop instilled in each affected eye 3 times a day for 7 days
  Interventions: Drug: Brinzolamide ophthalmic suspension, 1%
- Brimonidine (Active Comparator): Brimonidine tartrate ophthalmic solution, 0.2%, 1 drop instilled in each affected eye 3 times a day for 7 days
  Interventions: Drug: Brimonidine tartrate ophthalmic solution, 0.2%

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
  Arms: Brinz/Brim
Drug: Brinzolamide ophthalmic suspension, 1%
  Arms: Brinzolamide
Drug: Brimonidine tartrate ophthalmic solution, 0.2%
  Arms: Brimonidine

SUMMARY:
The purpose of this study was to describe the ocular discomfort immediately upon instillation of Brinzolamide 1%/Brimonidine 0.2% Tartrate Ophthalmic Suspension, Brinzolamide 1% Ophthalmic Suspension, and Brimonidine Tartrate 0.2% Ophthalmic Solution in subjects with open-angle glaucoma and/or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Diagnosis of open-angle glaucoma or ocular hypertension
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential if pregnant, lactating, or not using highly effective birth control measures.
* Severe central vision loss in either eye.
* Any chronic or recurrent inflammatory eye disease.
* Ocular trauma within the preceding 6 months.
* Ocular infection or ocular inflammation within the preceding 3 months.
* Best-corrected visual acuity score worse than 55 letters using the Early Treatment Diabetic Retinopathy Study chart.
* Any intraocular surgery within the preceding 6 months.
* Any ocular laser surgery within the preceding 3 months.
* History or current evidence of severe illness or any other conditions which would make the subject, in the opinion of the Investigator, unsuitable for the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravaughn Williams, OD, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 investigational centers in the United States.
Pre-assignment Details: Of the 103 enrolled, 2 subjects did not meet inclusion/exclusion criteria and were exited from the study as screen failures prior to randomization. This reporting group includes all randomized subjects (101).
Period: Overall Study
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine
Started | 33 | 34 | 34
Completed | 33 | 34 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine | Total
Number analyzed (Participants) | 33 | 34 | 34 | 101
Age, Customized [Number; unit: participants]
  18 to 64 years | 8 | 12 | 11 | 31
  ≥65 years | 25 | 22 | 23 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 23 | 66
  Male | 13 | 11 | 11 | 35
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 34 | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Discomfort Score
Description: Ocular discomfort was assessed by the subject immediately following the 8 AM instillation of study drug and rated on a 5-point scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe), and 4 (very severe).
Time Frame: Week 1
Population: Intent-to-Treat (ITT): All subjects who received study medication and had at least 1 scheduled on-therapy visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine
Number analyzed (Participants) | 33 | 34 | 34
Units on a scale | 0.8 (0.9) | 0.4 (0.6) | 0.3 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all subjects who were exposed to study medication.
Description: An adverse event was defined as any untoward medical occurrence in a subject administered a study medication, regardless of whether or not the event had a causal relationship with the medication. Adverse events were obtained as solicited comments from the subjects and as observations by the Investigator as outlined in the study protocol.
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 5/33 | 7/34 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=33) | Brinzolamide (N=34) | Brimonidine (N=34)
Vision blurred (Eye disorders) | 2 | 4 | 0
Eye irritation (Eye disorders) | 2 | 3 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.